CLINICAL TRIAL: NCT04820517
Title: The Effect of Roy Adaptation Model Based Strengthening Program Applied to Nursing Students on Social Media Addiction
Brief Title: Roy Adaptation Model Based Strengthening Program and Social Media Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Zeliha YAMAN, Principal Investigator, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Social Media Addiction
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Social Media Addiction
Keywords: Social media addiction; Empowerment; Nursing; Roy Adaptation Model
MeSH Terms: conditions — Internet Addiction Disorder; Empowerment

STUDY DESIGN:
Intervention Model Description: This study is pretest posttest randomized controlled clinical trial. The universe of this study was composed of 411 nursing students studying at Mersin University's faculty of nursing.The data were collected using the Bergen Social Media Addiction Scale from 384 nursing students who accepted to participate in the study between 09 January 2020 - 09 March 2020.From the scale developed by Andresan et al in 2017 and adapted to Turkish by Demirci in 2019, 110 nursing students who scored 3 or more out of at least 4 out of 6 items or scored 18 or more out of the total score constituted the sample of the study.110 nursing students were assigned to the experimental and control groups (55 experimental and 55 control groups) by block randomization.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The Roy Adaptation Model Based Empowerment Program, which consists of 12 sessions that will create awareness of social media and its effects in students and contribute to students gaining and maintaining a healthy lifestyle by providing controlled and purposeful use of social media with behavioral change, will be held with online group sessions for 12 weeks to the students in the experimental group. .
  Interventions: Other: Roy Adaptation Model Based Strengthening Program
- Control Group (No Intervention): No intervention will be made to the students in the control group. When the research is completed, student nurses in the control group will be informed about social media addiction and its effects.

INTERVENTIONS:
Other: Roy Adaptation Model Based Strengthening Program — Applications included in the strengthening program sessions:
  * Awareness study on social media addiction and its effects
  * Awareness work on the correct and effective use of leisure time
  * As a result of social media addiction, within the scope of Roy Adaptation Model, scenario sharing and problem solving process related to the problems arising in the fields of physical, group identity - self, role and interdependence
  * Awareness work on recognizing and managing emotions
  * Relaxation and Breathing Exercise in Emotion Management
  Arms: Experimental Group

SUMMARY:
In this pretest-posttest, randomized controlled study, the effect of the empowerment program developed based on Roy Adaptation on the healthy lifestyle behaviors, self-esteem and social media addiction of nursing students will be examined. The hypothesis of this study is that the empowerment program based on Roy Adaptation Model reduces Social Media Addiction, increases Healthy Lifestyle Behaviors and Self-Esteem.

DETAILED DESCRIPTION:
The universe of this study was composed of 411 nursing students studying at Mersin University's faculty of nursing.The data were collected using the Bergen Social Media Addiction Scale from 384 nursing students who accepted to participate in the study between 09 January 2020 - 09 March 2020.From the scale developed by Andresan et al in 2017 and adapted to Turkish by Demirci in 2019, 110 nursing students who scored 3 or more out of at least 4 out of 6 items or scored 18 or more out of the total score constituted the sample of the study.110 nursing students were assigned to the experimental and control groups (55 experimental and 55 control groups) by block randomization.7 separate focus group sessions were held online between 01 September 2020 - 01 October 2020 with 55 student nurses in the experimental group. Using the literature and data obtained from the first stage of the study (analysis of focus group sessions), a strengthening program based on the Roy Adaptation Model was made.The necessary corrections and additions were made to the program by obtaining expert opinions from field experts regarding the program created. Empowerment program based on Roy Adaptation Model will be applied to 55 student nurses in the experimental group between 01 February 2021 - 01 May 2021 through online group sessions. The Bergen Social Media Addiction Scale, Rosenberg Self-Esteem Scale and Healthy Lifestyle Behaviors Scale, which were applied as a pre-test in the first session of the application, will be applied as a post-test in the 12th session.

ELIGIBILITY:
Inclusion Criteria:

* agreeing to participate in research
* students who score 3 or more out of at least 4 out of 6 items or score 18 or more out of the total score in the Bergen Social Media Addiction Scale.

Exclusion Criteria:

* who do not agree to participate in the research
* students who scored 3 or less from at least 3 out of 6 items in the Bergen Social Media Addiction Scale, or who scored 17 or less out of the total score

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Addiction level changed using Bergen Social Media Addiction Scale in | Change from before implementation and 12th week of practice.
  The scale is answered according to five-point Likert-type grading ranging from (1) very rare to (5) very frequent. The total score of the scale varies between 6-30. As the scores obtained from the scale increase, the level of social media addiction also increases.

SECONDARY OUTCOMES:
Healthy lifestyle evaluated using the Healthy Lifestyle Behaviors Scale | Change from before implementation and 12th week of practice.
  The rating is in the form of a 4-point Likert. It is accepted as never (1), sometimes (2), often (3), regularly (4). For the whole scale, the lowest score is 52, the highest score is 208. While the maximum points that can be obtained from the sub-dimensions of health responsibility, nutrition, spiritual development and interpersonal relations are 36, the minimum points are 9. While the maximum scores from physical activity and stress management sub-dimensions are 32, the minimum scores are 8. The high score obtained from the Healthy Lifestyle Behaviors Scale indicates that the individual has more positive health behaviors in his life.

OTHER OUTCOMES:
Self-esteem evaluated using the Rosenberg Self-Esteem Inventory | Change from before implementation and 12th week of practice.
  The score obtained from the scale varies between 0-30. The higher the score, the higher the self-esteem. Thirty points are considered as self-esteem at the maximum level, 15-25 as normal self-esteem, and below 15 points as decreased self-esteem.

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yaman Z, Yilmaz M. The effect of the programme based on Roy adaptation model on social media addiction, healthy lifestyle and self-esteem of nursing students. Int J Nurs Pract. 2024 Aug;30(4):e13218. doi: 10.1111/ijn.13218. Epub 2023 Nov 17. PMID 37974502